CLINICAL TRIAL: NCT04020224
Title: A Randomized, Controlled, Phase I Clinical Trial to Assess the Safety of Whole Blood Treated With Amustaline (S-303) and Glutathione (GSH), a Pathogen Reduction System, in Anemic Patients
Brief Title: INTERCEPT Safety Evaluation on Whole Blood
Acronym: POINT1africa
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Sponsor's decision
Sponsor: Swiss Transfusion SRC (Other)
Collaborators: Cerus Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 1702005
Record Dates: First submitted 2019-07-09; First posted 2019-07-15 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Safety Issues
Keywords: anemia; transfusion; pathogen inactivation; pathogen reduction; low-resource; sub-saharan africa; transfusion-transmitted infection; whole blood
MeSH Terms: conditions — Anemia; Transfusion Reaction

STUDY DESIGN:
Intervention Model Description: 10 patients in the Test arm 10 patient in the Control arm
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment with pathogen reduced whole blood (Experimental): Subjects will receive one amustaline/GSH treated whole blood product.
  Interventions: Device: Amustaline/GSH pathogen reduction technology
- Treatment with Standard of Care (Active Comparator): Subjects will receive the Standard of Care (SOC), either one red blood cell (RBC) component or one whole blood product
  Interventions: Device: Standard of Care

INTERVENTIONS:
Device: Amustaline/GSH pathogen reduction technology — Whole blood treated with pathogen reduction technology
  Arms: Treatment with pathogen reduced whole blood
Device: Standard of Care — Red Blood Cell Component or whole blood
  Arms: Treatment with Standard of Care

SUMMARY:
The pathogen reduction system for whole blood using amustaline (S-303) and glutathione (GSH) hast a potential to decrease transfusion-transmitted infection. There is a scientific basis to hypothesize, that cells containing DNA and RNA such as bacteria, viruses and parasites that could be present in blood collected from asymptomatic infected donors are inactivated in the treated whole blood and therefore reduce the risk of transfusion-transmitted infections.

The aim of the study is to assess the safety of whole blood treated with amustaline and glutathione and transfused in patients with anemia.

This is a first-in-human-subjects study. Whole blood (WB) products treated with the amustaline (S-303) and glutathione (GSH) pathogen reduction technology have not been evaluated in human beings. However, red blood cells concentrates treated with amustaline and GSH have been evaluated in multiple clinical studies.

The study described in this protocol is a randomized, controlled, open-label Phase I clinical trial.

20 patients will be randomized into either the Test or Control arm in a ratio of 1:1.

10 patients assigned to the Test arm will receive one amustaline/GSH treated whole blood product.

10 patients assigned to the Control arm will receive the Standard of Care (SOC), either one red blood cell (RBC) component or one whole blood product.

DETAILED DESCRIPTION:
Screening:

All potentially eligible patients at the participating institution will be approached for study consent prior to study transfusion. Enrolled patients will also be asked for consent to the storage of their samples for future research on Transfusion Transmitted Infections (TTI). Illiterate patients can be consented by an impartial witness (see section 2.7).

Patients who consent to the study will be assigned a study identification (ID) number and undergo screening.

Screening data collection and procedures will include: Demographics (age, sex), vital signs, height, weight, indication for anticipated transfusion, medical history including history of bleeding and transfusion and concomitant medications. A physical examination, including skin inspection, will be performed. Blood samples will be drawn for a hematological panel (including complete blood count, blood chemistry, blood type, coagulation (aPTT, PT and/or INR) and pregnancy test (if applicable). Immunohematology tests will be performed on a patient's sample at the blood center. This includes a Direct Antibody Test (DAT), immune reactivity to RBCs that have been processed with amustaline and glutathione, red cell alloantibody screen (Indirect Antibody Test (IAT) / Indirect Coombs).

Blood samples (pre/post-treatment) for future research on TTIs will be archived in a biobank of the Institut Pasteur de Côte d'Ivoire (IPCI) (see section 9.3.3.11).

Randomization:

After successful screening, eligible patients will be assigned to a treatment arm by randomization. Randomization will be performed in the blood center by sequentially selecting a randomization envelope starting with the lowest number (e.g., 1 for the first eligible subject in ascending order up to envelope number 20 for the 20th subject).

The ratio of patients assigned to the Test and Control group will be 1:1. Each subject will receive a Test product or an untreated product based on existing SOC. The assigned blood product number must be noted on the randomization assignment envelope and on the release form. The product number will also be entered into the case report form (CRF).

The replacement strategy in this Phase I clinical trial is based on the aim to reach twenty evaluable patients. "Evaluable patients" is defined as those patients who are randomized and receive any study transfusion.

If a randomized subject withdraws or is withdrawn from the study prior to the administration of any study transfusion, or does not receive any study transfusion through 7-days post-randomization, this subject will be replaced by the next eligible subject using the same randomization envelope. If a randomized subject receives a conventional (untreated) blood transfusion prior to study transfusion, the patient will be replaced as described above.

All patients who received at least one investigational product will be included in the analysis (i.e., group of 20 evaluable patients) and followed through the final Day 58 study visit).

All used and unused randomization envelopes will be kept in the Site File for reconciliation.

Pre-transfusion visit:

Vital signs, weight, skin inspection will be performed, hemoglobin will be assessed, and urine samples will be taken for detection of blood in urine. If the patient consents to future research on TTI, a sample will be drawn and sent to the archival biobank.

Treatment:

Patients will be transfused with one investigational product or SOC on Day 1. In case he or she requires further transfusion support to treat anemia, enrolled patients may be treated with a second study transfusion. A patient who requires a second blood component within the first 24 hours will receive a second treatment, if available, with an investigational product from the assigned treatment arm. This patient will be included into the analysis of evaluable patients and followed up to Day 58, the final study visit. If the patient requires further transfusions (third transfusion etc.) it will be SOC.

Post-transfusion visit(s):

Patients will be hospitalized for 24 hours after each study transfusion to allow close monitoring and data collection uniquely for the study purpose since their condition would allow an outpatient treatment. 3 hours and 6 hours after initiating each study transfusion vital signs and skin inspection will be performed.

24-hours post-transfusion vital signs, urine dipstick, concomitant medication/intervention will be assessed, laboratory blood samples for hemoglobin, coagulation assays (aPTT, PT and/or INR) and potassium and a sample for determination of residual S-300 will be taken.

If a subject consented to future research on TTI, a second blood sample (post-transfusion) will be collected and archived in the biobank.

In case clinical symptoms of transfusion-related bacterial contamination occur, a blood sample will be collected during the post-transfusion period and microbiological analysis will be performed according to standard procedures in the IPCI. Those patients will be treated according to SOC.

Interim Safety Follow-up visit Day 14 days (+/-3 days) after last study transfusion: adverse event and and concomitant medication.

Final Safety Follow-up visit Day 28 days (+/-3 days) after last study transfusion:

At day 28 (+/-3 days) a physical examination, vitals, urine dipstick and blood samples will be collected for laboratory analysis of safety variables (e.g., complete blood count, coagulation) and urine dipstick.

All Adverse Events (AE), Transfusion Reactions (TR) and unanticipated adverse device effects will be reviewed and recorded for the period from the first study transfusion through Day 28 after the last study transfusion.

The Investigators will assess each AE for relation to the study transfusion. Available clinical diagnostic tools will be used to rule out unrelated AEs and to classify possible, probable and certain TRs using Swissmedic causality definitions.

Final study visit on Day 58 (+/-7 days) after last study transfusion) At the final study visit, the immune reactivity of patient serum to RBCs treated with amustaline/GSH for patients in the test arm and a DAT test for all patients will be performed.

Serious Adverse Events (SAEs) will be reviewed and recorded for the full study period from transfusion through to Day 28, which is the day of the final safety follow-up study visit.

The Investigators will assess each SAE for relation to the study transfusion. As SAEs will be further evaluated as possible transfusion reactions. SAEs that are determined to be possibly, probably or certainly related to the transfusion will be classified as TRs.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must be18 years of age or older;
2. Patients should have poorly tolerated anemia with a hemoglobin level greater than or equal to 5.0 g/dl and less than or equal to 7.0 g/dl. At the discretion of the investigator, inclusion is possible at a hemoglobin level greater than 7.0 g/dl if the criteria in the current local guidelines are met.
3. Patients must sign the study's informed consent form prior to initiation of any study-specific procedure / treatment. Enrolled patients may give additional consent for specimens collected during this study to be used for future research on TTIs. Patients may participate in the main trial and decline collection of specimens for future research.
4. Patients must agree to be hospitalized for a maximum of 72 hours after initiation of a study transfusion;
5. Female patients of childbearing potential must:

   1. have a negative serum pregnancy test within 72 hours prior to receiving the first study blood to rule out pregnancy, and;
   2. use at least one method of birth control that results in a low failure rate (i.e., less than 1% per year) when used consistently and correctly. These include combined oral contraceptives, implants, injectable, some intrauterine devices, sexual abstinence or vasectomized partner. The selected method must be used for the duration of study participation that means from day 1 (day of initiation of study transfusion) until day 58 (Final Study Visit).

Exclusion criteria:

The presence of any one of the following exclusion criteria will lead to exclusion:

1. Patients with blood group AB and blood group O Rhesus negative (due to concern of limited supply).
2. Positive antibody screening reaction specific to red blood cells treated with amustaline and glutathione (GSH).
3. Positive red cell alloantibody screening (IAT) / presence of red cell antibodies;
4. Patient has ongoing clinical-significant bleeding described as grade 2 or more according to the U.S. National Cancer Institute's CTCAE v5.0 severity grading scale.
5. Lifelong history of major bleeding due to congenital or acquired coagulopathy.
6. History of thrombosis or thromboembolic events.
7. Blood in feces or hemoglobinuria in the last 30 days.
8. Pre-transfusion thrombocyte counts of < than 50 Giga/l (x109).
9. Oral, intravenous or sub-cutaneous prophylactic or therapeutic anticoagulants.
10. Central body temperature increase of ≥2°C within 24 hours before transfusion.
11. Clinical signs of ongoing sepsis including fever >39°C with signs of a systemic, inflammatory response.
12. Abnormal activated partial thromboplastin time (aPTT) and/or abnormal prothrombin time (PT) or INR laboratory results
13. Transfusion of a blood product within 2 weeks prior to enrollment.
14. Abnormal total bilirubin (≤ 2 x upper limit of normal) levels and/or clinical signs of jaundice.
15. Sickle cell anemia.
16. Malignant cancer patients having received chemotherapy within 12 months.
17. Patients in need of multiple RBC or WB transfusions in the first 24 hours according to the investigator's judgment (i.e., more than one product).
18. Pregnant or breast-feeding.
19. Inability to comply with the protocol in the opinion of the investigator.
20. Participation in any other type of clinical study, either concurrently or within the previous 30 days, including: investigational blood products, nutrition, pharmacologic agents or imaging materials, including dyes, investigational surgical techniques, or devices. Studies of psychology or socioeconomic issues are not grounds for exclusion.
21. Participation on not more than two research studies per year.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-01 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Severe Transfusion Reactions | 24 hours
  The primary safety outcome will be assessed by the occurrence of transfusion reactions >= grade 2 according to the Swissmedic transfusion reaction grading and causality criteria (Appendix 1: Swissmedic Classification and Analysis of Transfusion related reactions ), during the first 24 hours following administration of each study transfusion, with probable, possible or certain causality to the transfused product.

SECONDARY OUTCOMES:
Adverse Events | 28 days (+/-3 days)
  All Adverse Events including transfusion reactions within 28 days (+/-3) after last study transfusion
Treatment-induced antibodies | 58 days (+/-7 days)
  Treatment-induced antibodies to amustaline/GSH treated RBCs within 58 (+/-7) days after last study transfusion.
Treatment-induced auto-antibodies | 58 days (+/-7 days)
  Treatment-induced auto-antibodies within 58 (+/-7) days after last study transfusion.
24 h post-transfusion hemoglobin | 24 hours
  Hemoglobin increment 24h post-transfusion adjusted by hemoglobin content transfused.

CONTACTS AND LOCATIONS:
Overall Officials: Soraya Amar, Dr, Principal Investigator — SwissTransfusion SRC

IPD SHARING:
Plan to Share IPD: No